CLINICAL TRIAL: NCT05875480
Title: Compare the Effects of Telerehabilitation and Conventional Rehabilitation After Artroscopic Meniscus Surgery
Brief Title: The Effectiveness of Telerehabilitation After Arthroscopic Meniscus Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Burcu Özdemir Kocabey, MSc, PhD(c), Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BahcesehirUniversitiy
Record Dates: First submitted 2023-04-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Telerehabilitation; Meniscus Tear; Physiotherapy; Rehabilitation; Postoperative
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- synchronized telerehabilitation group (Experimental): Patients in the synchronized telerehabilitation group had taken real time videoconferencing rehabilitation by physiotherapist 2 times a week, during 4 weeks.
  Interventions: Procedure: synchronized telerehabilitation
- asynchronized telerehabilitation group (Experimental): Patients in the asynchronized telerehabilitation group had done the postoperative rehabilitation with exercise videos via application.
  Interventions: Procedure: asynchronized telerehabilitation
- supervized conventional rehabilitation group (Active Comparator): Patients in the supervised physiotherapy group had taken their rehabilitation sessions in the physiotherapy department of the hospital twice a week, during 4 weeks.
  Interventions: Procedure: supervised (face to face) rehabilitation

INTERVENTIONS:
Procedure: synchronized telerehabilitation — In the synchronized telerehabilitation group, the exercise program of the first 2 weeks was submitted via Albert Health Assistant application and patients were asked to do these exercises regularly during this process. after 2 weeks, they were treated 2 days a week until the 6th week by meeting with the physiotherapist in real time via the Albert Health Assistant application. In the remaining days, they were asked to follow the exercise videos uploaded to the Albert system, it will be checked whether they have done the daily exercises, and a daily reminder message will be sent through the system.
  Arms: synchronized telerehabilitation group
Procedure: asynchronized telerehabilitation — The exercise program for the asynchronized telerehabilitation group will be uploaded to the Albert Health Assistant in the form of 2-week programs in video form from the first Day. Whether the patients apply these videos on a daily basis will be checked through the system, a message reminding the daily routine exercise program will be sent through the system.
  Arms: asynchronized telerehabilitation group
Procedure: supervised (face to face) rehabilitation — In the supervised physiotherapy group, the exercise program of the first 2 weeks was submitted via Albert Health Assistant application and patients were asked to do these exercises regularly during this process. After 2 weeks, they attended the rehabilitation program in the physical therapy department of the hospital accompanied by a physiotherapist, starting from the 14th postoperative day, 2 days a week until the 6th week. The ROM, pain, functional and general health evaluations of the patients in this group were carried out on the online platform. In addition, on the days when they did not come to treatment, their daily routine exercises were followed through the Albert system.
  Arms: supervized conventional rehabilitation group

SUMMARY:
This study was performed on 42 patients, who underwent arthroscopic meniscus repair surgery in the Orthopedics and Traumatology Department of Acıbadem Maslak Hospital. 42 patients randomly assigned to 14 synchronized telerehabilitation, 14 asynchronous telerehabilitation, 14 conventional physiotherapy groups and included in the study. The evaluation form created for the provision of demographic information are used.

Primary outcome measures are muscle strength, range of motion (ROM) and pain intensity.

Secondary outcome measures are general health profile and functional status assessment of the knee joint .

Evaluation methods: All evaluations were performed in the preoperative period, 10. day, 6. week and 6. month postoperatively. ROM and pain measurements repeated every week during the 6-week rehabilitation process.

Pain, general health profile and functional status assessment of the knee joint were assessed via a telerehabilitation application, Albert Health Assistant.

Postoperative first day, the 14-day exercise program was taught to all patients practically and was given as a brochure.

Patients in the synchronized telerehabilitation group started physiotherapy postoperative 14. day, met with the physiotherapist in real time via the Albert Health Assistant application and they were treated 2 days a week until 6. week. In the remaining days, they asked to follow the exercise videos uploaded to the Albert system, it was checked whether they are doing daily exercises, and a daily reminder message was sent via the system.

The exercise program for the asynchronous telerehabilitation group was uploaded to the Albert Health Assistant as a video from the 14th day in the form of 2-week programs. It was checked over the system whether the patients apply these videos on a daily basis, and a message reminding the daily routine exercise program was sent through the system.

Patients in the supervised physiotherapy group started to take supervized rehabilitation after 10-14 days postoperatively, 2 times a week until 6th week postoperatively in Maslak Acıbadem Hospital Orthopedics and Traumatology Department. ROM, Pain, functional and general health evaluations of the patients in this group were performed on the online platform. In addition, daily routine exercises will be followed over the Albert system on the days they do not come for treatment.

DETAILED DESCRIPTION:
Albert Health Assistant is an artificial intelligence-based digital health assistant that helps patients with their treatment. Albert is a healthcare assistant who ensures that patients take their medications at the right dose and at the right time, helps them with treatment compliance, and allows patient relatives and the attending physician to closely monitor the patient's treatment. Albert is a mobile software and sensitive qualified personal health data (patient information) are stored in accordance with the personal data protection law. n this process, which will be created with the Albert treatment tracking system, the following data types can be tracked remotely.

Primary Outcome measures:

Joint Range of Motion (ROM) measurement: Passive hyperextension angles was measured with the knee in active flexion and prone position (with gravity effect).

Joint range of motion measurement was performed with Dr Goniometer, a smartphone app. With this application, a photograph was taken from the patient at the maximum flexion angle that he can perform, and the measurement was made by placing markers on the reference points determined on the photograph. This application is found to be reliable in measuring the knee joint angle.

Muscle strength measurement: It was performed with a Lafayette hand dynamometer. The maximal isometric muscle strength of the hamstring and quadriceps muscles were tested 3 times and the average of 3 measurements were taken. The contraction time is 5 seconds, the rest time is 10 seconds, there was a resting period of 2 minutes in the tests between the two muscles. Measurements will be performed by placing the dynamometer on the distal 1/3 of the thigh while the prone knee is in the 45 degree flexion position.

Pain assessment: Visual Pain Scale (VAS) was used. VAS is a scale between 0-10 points. 0 corresponds to no pain, 10 corresponds to unbearable pain. It is a validated scale in which the patient self-assesses his pain at the time of evaluation.

Secondary Outcomes:

General Health profile measurement: It will was performed using the PROMIS 29 Health Profile Questionnaire. The Patient-Reported Outcomes Measurement Information System (PROMIS) is a general health scale created by the National Institutes of Health, in which the patient can self-report to assess functioning and well-being in the physical, mental and social areas of health.

IKDC subjective knee form: The IKDC (International Knee Documentation Committee) subjective knee form is designed to measure symptoms and limitations in function and sports activity for various knee conditions, including ligament, meniscus, and cartilage injuries, as well as patellofemoral pain.

ELIGIBILITY:
Inclusion Criteria:

* In the 18-50 age range,
* repairable, stable, longitudinal vertical longitudinal or bucket handle meniscus lesion,
* persons who volunteered to participate in the study

Exclusion Criteria:

* Meniscus root repair,
* Associated anterior cruciate ligament reconstruction,
* Other ligament injuries or laxity,
* Cartilage lesion larger than 2 cm² in size and more than half the thickness of the cartilage (International Society for Cartilage Research [ICRS] grade 3 or 4),
* previous meniscus or ligament surgery,
* presence of congenital lower extremity deformity,
* hip and ankle joint pathologies,
* the presence of systemic diseases affecting the joints such as rheumatoid arthritis
* lack of ability to follow the established rehabilitation program

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 6 minutes
  Muscle strength measurements were made with a Lafayette hand dynamometer. The maximal isometric muscle strength of the hamstring and quadriceps muscles was tested 3 times and the average of 3 measurements was taken. The contraction time was 5 seconds, the rest time was 10 seconds, and a 2-minute rest period was given in the tests between the two muscles. Measurements were made with the prone knee in the 45 degree flexion position, with the dynamometer placed on the distal 1/3 of the thigh.
Range of motion of knee joint | 1-2 minutes
  Range of motion measurement was performed every week between the 1st-6th weeks postoperatively and once in the 6th month. Passive hyperextension angles of the knee were measured in active flexion and prone position (with the effect of gravity).
  Joint range of motion measurement was performed with Dr Goniometer, a smartphone application. With this application, a photograph was taken from the patient at the maximum flexion angle that he could achieve, and the measurement was made by placing markers on the reference points determined on the photograph.
Pain intensity | less than 1 minute
  Visual Pain Scale (VAS) was used. VAS is a scale between 0-10 points. 0 corresponds to no pain, 10 corresponds to unbearable pain. It is a validated scale in which the patient self-assesses their pain at the time of assessment.

SECONDARY OUTCOMES:
Functional knee assessment | 5-6 minutes
  It was evaluated using the IKDC (International Knee Documentation Committee) subjective knee form. This form is designed to measure symptoms and limitations in function and sporting activity for a variety of knee conditions, including ligament, meniscus and cartilage injuries, as well as patellofemoral pain.
General health profile | 5-6 minutes
  It was conducted using the Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) Health Profile Questionnaire. PROMIS -29 is a general health scale created by the National Institutes of Health, where the patient can self-report to assess functioning and well-being in the physical, mental and social areas of health. It includes 28 items from seven PROMIS domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities) and a single item on pain intensity.Each item has five response options (values 1 to 5), except for the pain intensity item which has eleven response options (values 0 to 10). A total raw score is computed for each domain as the sum of the response to each question within the domain, leading to seven domain scores, each from 4 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Dilber Coşkunsu, Assoc. Prof., Study Director — Fenerbahçe University
Locations (1):
- Maslak Acıbadem Hospital, Istanbul, Turkey (Türkiye)